CLINICAL TRIAL: NCT01370317
Title: Multiple Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of MK-1029 or Placebo in Patients With Mild to Moderate Asthma
Brief Title: Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MK-1029 in Participants With Mild to Moderate Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1029-006; MK-1029-006 (Other: Merck Protocol Number)
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-1029 (Experimental)
  Interventions: Drug: MK-1029
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo for MK-1029

INTERVENTIONS:
Drug: MK-1029 — Five (5) X 100 mg capsules, orally, once daily for 28 days
  Arms: MK-1029
Drug: Placebo for MK-1029 — Five (5) X 100 mg capsules, orally, once daily for 28 days
  Arms: Placebo

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics (PK) of multiple dose treatment with MK-1029 in adults with mild to moderate persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* If female, must be of non-childbearing potential
* Have a history of mild to moderate asthma for at least 6 months
* Other than asthma, in general good health
* Able to perform reproducible pulmonary function testing
* Is a nonsmoker and/or has not used nicotine or nicotine-containing products for at least 12 months
* Have body mass index (BMI) ≥17 kg/m^2, but ≤35 kg/m^2

Exclusion Criteria:

* Demonstrate a decrease in absolute forced expiratory volume in 1 second (FEV1) of >20% from the Screening Visit to the Baseline Visit
* Experience a decrease in AM or PM peak expiratory flow (PEF) below the Stability Limit on any 2 consecutive days prior to the Baseline Visit
* Require the use of >8 inhalations per day of short-acting beta2-agonist metered dose inhaler (MDI) or >2 nebulized treatments per day of 2.5 mg albuterol, on any 2 consecutive days from the Screening Visit up to the Baseline Visit
* Experience an exacerbation defined as a clinical deterioration of asthma, as judged by the clinical investigator, that results in emergency treatment, hospitalization due to asthma, or treatment with additional, excluded medication (other than short-acting beta agonists [SABA]) at any time from the Screening Visit up to the Baseline Visit
* Have been hospitalized for treatment of asthma or required oral corticosteroids for treatment of asthma within the past 6 months, or has ever required ventilator support for respiratory failure secondary to asthma
* Require the chronic use of high-dose inhaled corticosteroids
* Have been diagnosed with chronic obstructive pulmonary disease (COPD) or any other clinically relevant lung disease, other than asthma
* Have a history of any illness that might confound the results of the study or poses additional risk to the participant
* Have had recent (within 4 weeks of first dose) or ongoing upper or lower respiratory tract infection
* Is nursing
* Have a history of significant multiple and/or severe allergies (including latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2011-12-27 (Actual); Study Completion 2011-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- United States (2):
  - Call for Information, Costa Mesa, California
  - Call for Information, Rolling Hills Estates, California
- Merck Sharp & Dohme, North Ryde, Australia
- Merck Sharp & Dohme (New Zealand) Ltd.,, Wellington, New Zealand
- MSD (Pty) LTD South Africa, Midrand, South Africa

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-1029: Participants received five 100 mg MK-1029 capsules, taken orally, once daily for 28 days.
- Placebo: Participants received five 100 mg placebo-matching MK-1029 capsules, taken orally, once daily for 28 days.
Period: Overall Study
Arm/Group | MK-1029 | Placebo
Started | 18 | 9
Completed | 17 | 8
Not Completed | 1 | 1
Not completed — Participant withdrew consent | 1 | 0
Not completed — Protocol deviation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-1029 | Placebo | Total
Number analyzed (Participants) | 18 | 9 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.4 (15.2) | 41.6 (13.5) | 40.8 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 11
  Male | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced One or More Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a study participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to 42 days after initial dose of study treatment
Population: All participants who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1029 | Placebo
Number analyzed (Participants) | 18 | 9
Participants | 9 | 3

2. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to 6 Hours (AUC0-6hr) of MK-1029
Description: Blood was collected on Day 1 and Day 28 at predose and 1, 2, 3, 4 and 6 hours postdose for determining the Cmax of MK-1026.
Time Frame: Day 1 and Day 28: Predose, 1, 2, 3, 4, and 6 hours postdose
Population: All participants who received study drug and had evaluable concentration values for AUC0-6 hours on Day 1 and Day 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | MK-1029
Number analyzed (Participants) | 16
ng*hr/mL
  Day 1: number analyzed (Participants) | 15
  Day 1 | 745 (104)
  Day 28: number analyzed (Participants) | 14
  Day 28 | 505 (275)

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MK-1029
Description: as for outcome 2
Time Frame: Day 1 and Day 28: Predose, 1, 2, 3, 4, and 6 hours postdose
Population: All participants who received study drug and had evaluable concentration values for Cmax on Day 1 and Day 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MK-1029
Number analyzed (Participants) | 16
ng/mL
  Day 1 | 295 (106)
  Day 28: number analyzed (Participants) | 14
  Day 28 | 167 (273)

4. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of MK-1029
Description: Blood was collected on Day 1 and Day 28 at predose and 1, 2, 3, 4 and 6 hours postdose for determining the Tmax of MK-1026.
Time Frame: Day 1 and Day 28: Predose, 1, 2, 3, 4, and 6 hours postdose
Population: All participants who received study drug and had evaluable concentration values for Tmax on Day 1 and Day 28
Measure: Median (Full Range); unit: Hours
Arm/Group | MK-1029
Number analyzed (Participants) | 16
Hours
  Day 1 | 2.00 [2.00 to 3.08]
  Day 28: number analyzed (Participants) | 14
  Day 28 | 3.00 [1.98 to 4.00]

5. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to An Adverse Event
Description: An AE is any untoward medical occurrence in a study participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to 28 days after initial dose of study treatment
Population: All participants who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1029 | Placebo
Number analyzed (Participants) | 18 | 9
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 42 days after initial dose of study treatment
Description: All participants who received at least one dose of study drug
Arm/Group | MK-1029 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/9
Other Adverse Events (participants affected / at risk) | 9/18 | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1029 (N=18) | Placebo (N=9)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Otitis media viral (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 2 (3) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Heat rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.